CLINICAL TRIAL: NCT01810224
Title: Graft Patency After FFR-guided Versus Angio-guided CABG: a Prospective, Multicenter, Multinational, Randomized (1:1) Controlled Trial
Brief Title: Graft Patency After FFR-guided Versus Angio-guided CABG (GRAFFITI) Trial
Acronym: GRAFFITI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Emanuele Barbato, Doctor, Onze Lieve Vrouw Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRAFFITI
Record Dates: First submitted 2013-03-09; First posted 2013-03-13 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angio-guided arm (Active Comparator): In this arm will be included the patient randomized to a Angiography-guided surgical revascularization strategy.
  Interventions: Procedure: Surgical revascularization
- FFR-guided arm (Experimental): In this arm will be included the patient randomized to a FFR-guided surgical revascularization strategy.
  Interventions: Procedure: Surgical revascularization

INTERVENTIONS:
Procedure: Surgical revascularization — The final intervention (surgical revascularization) will be the same for both arms.

SUMMARY:
This is prospective, randomized, multicenter, multinational, randomized (1:1) study. The aim of this study is to assess the importance of functional assessment of coronary artery disease prior to bypass surgery. In particular, an FFR-guided strategy will be compared to the traditional Angio-guided strategy in the guidance of surgical revascularization by aorto-coronary bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina, unstable angina or NSTEMI candidate to CABG
* Significant LAD and/or LM lesion - proved by FFR or Angiography AND
* At least one more, angiographycally intermediate lesion

Exclusion Criteria:

* Significant valvular disease with indication to surgical replacement
* Severe left ventricular dysfunction (EF<35%)
* Acute STEMI
* Atrial fibrillation, if Maze procedure is planned

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Rate of occluded bypass grafts | 1 year

SECONDARY OUTCOMES:
a) Lenght of hospital stay; b) Changes in surgical strategy: i.e. open-chest surgery vs. mini-thoracotomy; extensive surgery versus minimal invasive approaches. | participants will be followed for the duration of hospital stay, an expected average of 3-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Barbato, MD, PhD, Principal Investigator — Cardiovascular Center Aalst, OLV Hospital, Aalst (Belgium)
Locations (3):
- Cardiovascular Center Aalst OLV Hospital, Aalst, Belgium
- Department of Internal Medicine and Cardiology, University Hospital Brno, Brno, Czechia
- Hungarian Institute of Cardiology, Budapest, Hungary

REFERENCES:
- [Derived] Toth GG, De Bruyne B, Kala P, Ribichini FL, Casselman F, Ramos R, Piroth Z, Fournier S, Piccoli A, Van Mieghem C, Penicka M, Mates M, Nemec P, Van Praet F, Stockman B, Degriek I, Barbato E. Graft patency after FFR-guided versus angiography-guided coronary artery bypass grafting: the GRAFFITI trial. EuroIntervention. 2019 Dec 6;15(11):e999-e1005. doi: 10.4244/EIJ-D-19-00463. PMID 31270037
- [Derived] Toth GG, De Bruyne B, Kala P, Ribichini FL, Casselman F, Ramos R, Piroth Z, Fournier S, Van Mieghem C, Penicka M, Mates M, Van Praet F, Degriek I, Barbato E. Study Design of the Graft Patency After FFR-Guided Versus Angiography-Guided CABG Trial (GRAFFITI). J Cardiovasc Transl Res. 2018 Aug;11(4):269-273. doi: 10.1007/s12265-018-9818-9. Epub 2018 Jul 19. PMID 30027499